CLINICAL TRIAL: NCT04263935
Title: Correlation Between Driver Gene Abnormalities and Clinicopathological Characteristics and Disease Prognosis in Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanyan Liu, Director, Henan Cancer Hospital
Other Study IDs: HNCH2019341
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma; Gene Abnormality
Keywords: Lymphoma; Driver Gene Abnormalities; Disease Prognosis
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Correlation Between Driver Gene Abnormalities and Clinicopathological Characteristics and Disease Prognosis in Lymphoma

DETAILED DESCRIPTION:
This trial is a prospective non-interventional observational study. The Chinese patients with lymphoma were included and the study data on driver gene abnormalities, demographic characteristics, clinicopathological characteristics and treatment were collected to evaluate the relevance of efficacy and disease prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as lymphoma (according to WHO 2017 classification criteria)
2. Life expectancy no less than 3 months
3. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Other malignant tumor history or active malignant tumor need be treated
2. Researchers determine unsuited to participate in this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Including demographic characteristics / clinical characteristics / pathological characteristics / treatment and efficacy evaluations.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of driver gene abnormalities | from the day of the first patient was included to the date of the end of this trial, assessed up to 36 months
  the incidence of driver gene abnormalities by fixed gene testing technology

SECONDARY OUTCOMES:
objective response rate | from the date of the first patient was included to the date of the end of this trial, assessed up to 36 months
  the total proportion of patients with complete response (CR) and partial response (PR)
5-year overall survival | from the date of the first patient was included to the date of the end of this trial, assessed up to 5 years
  from the date of first patient was included to the date of death by any cause
Clinicopathological Characteristics | from the date of the first patient was included to the date of the end of this trial, assessed up to 36 months
  study data on clinicopathological characteristics related to incidence of driver gene abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No